CLINICAL TRIAL: NCT02977676
Title: Ventilator-Associated Events: Prevalence, Outcome and Preventability
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, Coordinator of ICU, Hospital Sao Domingos
Other Study IDs: CONEP 1.449.854
Record Dates: First submitted 2016-11-20; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Ventilator-Associated Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to determine the prevalence of ventilator-associated events (VAE). To analyze the patients profile, morbidity and mortality compared to patients who did not develope VAE. The preventability of VAE will be assessed by comparing the percentage of adherence to the bundle of preventive measures among patients who developed and did not develope VAE.

DETAILED DESCRIPTION:
This is a retrospective analysis of prospectively collected data, approved by the Research Ethics Committee of Hospital Sao Domingos. The need for informed consent was waived.

Included were all patients admitted to a surgical (13 beds) and medical (32 beds) of a tertiary hospital over a 3-year period (February 2013 to January 2016), aged above 18 years and submitted to mechanical ventilation for at least 4 days.

At admission and daily the following data were collected: head of bed elevation, daily interruption of sedation, gastric ulcer prevention, Thromboembolism prophylaxis, aspiration of subglottic secretions, oral care with chlorhexidine gluconate and monitoring of endotracheal tube cuff pressure.

Identification of VAE, Ventilator-associated condition (VAC), Infectious condition associated to mechanical ventilation (IVAC) and ventilator-associated pneumonia possible and probable followed definition criteria of the National Healthcare Safety Network / Center for Disease Control and Prevention.

The percentage of adherence to the bundle of preventive measures of VAE prevention was registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to a medical and a surgical ICUs over a 3-year period aged above 18 years and submitted to mechanical ventilation for at least 4 days.

Exclusion Criteria:

* Patients aged bellow 18 years and those that remained under mechanical ventilation less than 4 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a medical and a surgical ICUs over a 3-year period aged above 18 years and submitted to mechanical ventilation for at least 4 days.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-02; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who developed ventilator-associated events | 1 year
All cause Mortality | 1 year

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 1 year
Percentage of adherence to the package of VAE preventive measures | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, MA, PhD, Principal Investigator — Hospital Sao Domingos